CLINICAL TRIAL: NCT02271217
Title: This is a Multi-center, Double-blind, Three Arm, Parallel Group, Placebo-controlled, Randomized Study Designed to Evaluate the Efficacy, Safety and Tolerability of Dalfampridine.
Brief Title: A Study to Evaluate the Efficacy and Safety of Two Dose Strengths of Dalfampridine Extended Release Tablets.
Acronym: MILESTONE℠
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DALF-PS-1016
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2017-09

CONDITIONS: Post-Ischemic Stroke
Keywords: Post stroke; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Subjects randomized 1:1:1 to receive either dalfampridine-ER 7.5mg, dalfampridine-ER 10mg, or matching placebo tablets taken twice daily 12 hours apart.
  Interventions: Drug: Placebo
- dalfampridine-ER 7.5 mg (Active Comparator): Subjects randomized 1:1:1 to receive either dalfampridine-ER 7.5mg, dalfampridine-ER 10mg, or matching placebo tablets taken twice daily 12 hours apart.
  Interventions: Drug: dalfampridine-ER 7.5mg
- dalfampridine-ER 10mg (Active Comparator): Subjects randomized 1:1:1 to receive either dalfampridine-ER 7.5mg, dalfampridine-ER 10mg, or matching placebo tablets taken twice daily 12 hours apart.
  Interventions: Drug: dalfampridine-ER 10mg

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: dalfampridine-ER 7.5mg
  Arms: dalfampridine-ER 7.5 mg
Drug: dalfampridine-ER 10mg
  Other Names: Ampyra
  Arms: dalfampridine-ER 10mg

SUMMARY:
The objective of this study is to determine the effect of two dose strengths of dalfampridine-Extended Release (ER) tablets, taken twice daily for 12 weeks, on stable walking deficits in subjects with post-ischemic stroke.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, three-arm, parallel-group study designed to evaluate the efficacy, safety, and tolerability of dalfampridine extended release (ER) tablets on chronic walking deficits in subjects with post-ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of a stable walking deficit due to an ischemic stroke, as judged by the Investigator, based on review of medical records and physical exam. Such deficit was not present prior to the stroke and cannot be attributed primarily to other conditions (e.g. chronic obstructive pulmonary disease, arthritis). Evidence of walking deficits is objectively supported by any one of the following findings on clinical examination:

  1. obvious slowness of movement assigned primarily to the stroke
  2. use of an assistive walking device such as a cane or walker
  3. Presence of movement pattern deviations such as stiff-legged gait, foot drop, hip hiking and hip circumduction
* Modified Rankin Scale score of 1 - 3, regardless of the cause(s) of the disability
* Sufficient ambulatory ability to independently complete the 2MinWT and 10MWT
* ≥ 6 months from occurrence of most recent stroke

Exclusion Criteria:

* Woman who is not surgically sterile or is less than 2 years postmenopausal, and does not agree to use a highly effective birth control method during the study and up to 3 months after the last dose of investigational product.
* Woman who is pregnant, breastfeeding, or planning to become pregnant
* History of seizures, except simple febrile seizures
* Moderate or severe renal impairment as defined by a calculated creatinine clearance of ≤ 50 mL/minute using the Cockcroft-Gault Equation
* Suicide attempt within 1 year prior to the Screening Visit, or severe suicidal ideation within 6 months prior to the Screening Visit, or subject is at significant risk of suicidal behavior in the opinion of the Investigator
* Previous use of AMPYRA, dalfampridine, fampridine or 4-aminopyridine (4-AP)
* Initiation of a serotonin reuptake inhibitor (SSRI) within 3 months prior to the Screening Visit, or any change in dosing regimen within 3 months prior to the Screening Visit
* Botulinum toxin use within 2 months prior to the Screening Visit
* Orthopedic surgical procedures in any of the extremities within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Roberts, MD, Study Director — Acorda Therapeutics
Locations (74):
- United States (70):
  - Acorda Site #117, Gilbert, Arizona
  - Acorda Site #109, Berkeley, California
  - Acorda Site #138, Long Beach, California
  - Acorda Site #105, Newport Beach, California
  - Acorda Site #170, Oceanside, California
  - Acorda Site #142, Pasadena, California
  - Acorda Site #153, Sacramento, California
  - Acorda Site #151, San Diego, California
  - Acorda Site #163, San Diego, California
  - Acorda Site #124, Colorado Springs, Colorado
  - Acorda Site #110, Danbury, Connecticut
  - Acorda Site #149, Fairfield, Connecticut
  - Acorda Site #130, Stamford, Connecticut
  - Acorda Site #115, Atlantis, Florida
  - Acorda Site #119, Deerfield Beach, Florida
  - Acorda Site #147, Gainesville, Florida
  - Acorda Site #128, Hialeah, Florida
  - Acorda Site #143, Jacksonville, Florida
  - Acorda Site #103, Miami, Florida
  - Acorda Site #133, Miami, Florida
  - Acorda Site #161, Naples, Florida
  - Acorda Site #145, Sunrise, Florida
  - Acorda Site #106, Tampa, Florida
  - Acorda Site #186, Atlanta, Georgia
  - Acorda Site #181, Kailua, Hawaii
  - Acorda Site #171, Chicago, Illinois
  - Acorda Site #148, Avon, Indiana
  - Acorda Site #188, Fort Wayne, Indiana
  - Acorda Site #156, Franklin, Indiana
  - Acorda Site #146, Lexington, Kentucky
  - Acorda Site #150, New Orleans, Louisiana
  - Acorda Site #175, Fulton, Maryland
  - Acorda Site #136, Boston, Massachusetts
  - Acorda Site #121, Boston, Massachusetts
  - Acorda Site #120, Worcester, Massachusetts
  - Acorda Site #164, Bingham Farms, Michigan
  - Acorda Site #127, Detroit, Michigan
  - Acorda Site #123, East Lansing, Michigan
  - Acorda Site #159, Grand Rapids, Michigan
  - Acorda Site #101, Kansas City, Missouri
  - Acorda Site #111, Great Falls, Montana
  - Acorda Site #140, Reno, Nevada
  - Acorda Site #131, New Brunswick, New Jersey
  - Acorda Site #177, Stratford, New Jersey
  - Acorda Site #172, New York, New York
  - Acorda Site #102, New York, New York
  - Acorda Site #179, Patchogue, New York
  - Acorda Site #114, White Plains, New York
  - Acorda Site #166, Chapel Hill, North Carolina
  - Acorda Site #167, Durham, North Carolina
  - Acorda Site #162, Mooresville, North Carolina
  - Acorda Site #154, Raleigh, North Carolina
  - Acorda Site #132, Winston-Salem, North Carolina
  - Acorda Site #187, Bellevue, Ohio
  - Acorda Site #160, Cleveland, Ohio
  - Acorda Site #137, Columbus, Ohio
  - Acorda Site #116, Dayton, Ohio
  - Acorda Site #152, Corvallis, Oregon
  - Acorda Site #168, Portland, Oregon
  - Acorda Site #126, Portland, Oregon
  - Acorda Site #158, Abington, Pennsylvania
  - Acorda Site #122, Philadelphia, Pennsylvania
  - Acorda Site #144, Providence, Rhode Island
  - Acorda Site #157, Memphis, Tennessee
  - Acorda Site #113, Dallas, Texas
  - Acorda Site #165, Dallas, Texas
  - Acorda Site #108, Houston, Texas
  - Acorda Site #182, Alexandria, Virginia
  - Acorda Site #176, Richmond, Virginia
  - Acorda Site #107, Spokane, Washington
- Canada (4):
  - Acorda Site #203, Fredericton, New Brunswick
  - Acorda Site #202, Halifax, Nova Scotia
  - Acorda Site #201, Greenfield Park, Quebec
  - Acorda Site #204, Montreal, Quebec

REFERENCES:
- [Derived] Page SJ, Kasner SE, Bockbrader M, Goldstein M, Finklestein SP, Ning M, El-Feky WH, Wilson CA, Roberts H; all of the investigators involved in the MILESTONE study. A double-blind, randomized, controlled study of two dose strengths of dalfampridine extended release on walking deficits in ischemic stroke. Restor Neurol Neurosci. 2020;38(4):301-309. doi: 10.3233/RNN-201009. PMID 32651338
- See also: Click here for potential enrollment or for more information about this study: DALF-PS-1016 — http://milestone.acordatrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects randomized 1:1:1 to receive either dalfampridine-ER 7.5mg, dalfampridine-ER 10mg, or matching placebo tablets taken twice daily 12 hours apart.
  Placebo
- Dalfampridine-ER 7.5 mg: Subjects randomized 1:1:1 to receive either dalfampridine-ER 7.5mg, dalfampridine-ER 10mg, or matching placebo tablets taken twice daily 12 hours apart.
  dalfampridine-ER 7.5mg
- Dalfampridine-ER 10mg: Subjects randomized 1:1:1 to receive either dalfampridine-ER 7.5mg, dalfampridine-ER 10mg, or matching placebo tablets taken twice daily 12 hours apart.
  dalfampridine-ER 10mg
Period: Overall Study
Arm/Group | Placebo | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10mg
Started | 126 | 126 | 125
Completed | 115 | 113 | 113
Not Completed | 11 | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10mg | Total
Number analyzed (Participants) | 126 | 126 | 125 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (11.68) | 61.7 (10.48) | 64.3 (10.01) | 62.9 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 51 | 46 | 136
  Male | 87 | 75 | 79 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 20 | 59
  Not Hispanic or Latino | 108 | 105 | 105 | 318
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 2 | 6
  Asian | 3 | 4 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 18 | 12 | 21 | 51
  White | 100 | 105 | 94 | 299
  More than one race | 2 | 4 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight at Screening [Mean (Standard Deviation); unit: kg] | 83.98 (14.914) | 82.43 (14.514) | 84.49 (14.771) | 83.63 (14.72)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Show at Least a 20% Improvement on the Two Minute Walk Test (2MinWT) at Week 12
Description: "The 2MinWT measures the distance a subject can walk in 2 minutes. Participants showing at Least a 20% Improvement on the 2MinWT at 12-weeks are considered "Responders".
Time Frame: Week 12
Population: Includes all randomized subjects who took at least one dose of double-blind study treatment, had at least one 2MinWT assessment during the placebo run-in period, and at least one 2MinWT assessment during the double-blind treatment period.
Measure: Number; unit: participants
Arm/Group | Placebo | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 126 | 121 | 121
participants
  Responder | 17 | 17 | 23
  Non-Responder | 97 | 96 | 90
  Missing | 12 | 8 | 8

2. Secondary Outcome: Change From Baseline on the Walking Impact Scale (Walk-12) at Week 12 (Key Secondary)
Description: The Walk-12 is a 12-question questionnaire that asks subjects to rate limitations of their mobility during the preceding two weeks on a 5-point scale (from 1= not at all to 5=extremely). For each visit, the Walk-12 score will be calculated by summing the 12 components and transforming into a scale with a range of 0 to 100. A higher score indicates a greater degree of limitation in walking. A negative change indicates an improvement in walking. 0 = no limitation in mobility to 100 extreme limitation in mobility.
  Walk-12 Score = 100 * [(Mean of the 12 items) - 1]/(5-1)
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10mg
Number analyzed (Participants) | 126 | 121 | 121
units on a scale | 45.40 (22.96) | 48.34 (25.43) | 49.26 (25.98)

ADVERSE EVENTS:
Description: Clinicaltrials.gov definition of Adverse Events is any " Adverse events that are not Serious Adverse Events." The adverse events summary results provided for this study include both Serious Adverse Events and other Adverse Events that are not Serious Adverse Events.
  Adverse Events are reporting on the Safety Population which includes all subjects who received at least one dose of double-blind study treatment.
Arm/Group | Placebo | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10mg
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126 | 0/122
Serious Adverse Events (participants affected / at risk) | 8/126 | 6/126 | 3/122
Other Adverse Events (participants affected / at risk) | 75/126 | 85/126 | 75/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=126) | Dalfampridine-ER 7.5 mg (N=126) | Dalfampridine-ER 10mg (N=122)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Convulstion (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Complex Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=126) | Dalfampridine-ER 7.5 mg (N=126) | Dalfampridine-ER 10mg (N=122)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Fatigue (General disorders) | 8 (8) | 4 (4) | 3 (3)
Gait Disturbance (General disorders) | 0 (0) | 6 (6) | 0 (0)
Asthenia (General disorders) | 0 (0) | 4 (4) | 0 (0)
Edema Peripheral (General disorders) | 1 (1) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 8 (8) | 11 (11)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 12 (12) | 13 (13)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 4 (4)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Blood Glucose Increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 5 (5)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 4 (4)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) — SOC/PT
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) — SOC/PT
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) — SOC/PT
Dizziness (Nervous system disorders) | 3 (3) | 10 (10) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 6 (6) | 2 (2)
Balance Disorder (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 5 (5) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.